CLINICAL TRIAL: NCT02316652
Title: Using Chemical Pocket Disinfection as an Adjunct to Non-surgical Maintenance Therapy of Inflamed Periodontal Pockets
Brief Title: Effect of Disinfective Solution as an Adjunct to Maintenance Therapy of Inflamed Periodontal Pockets
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped and was not completed
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0636-13-FB
Record Dates: First submitted 2014-12-08; First posted 2014-12-15 (Estimated); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing; Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy sites (No Intervention): Healthy sites with no inflammation; observational only
- Scaling and root planing sites (Placebo Comparator): Inflamed pocket receiving mechanical instrumentation
  Interventions: Procedure: Scaling and root planing
- Scaling and root planing with solution (Active Comparator): Inflamed pocket receiving mechanical instrumentation with sodium hypochlorite solution
  Interventions: Procedure: Scaling and root planing with solution

INTERVENTIONS:
Procedure: Scaling and root planing — Mechanical instrumentation
  Arms: Scaling and root planing sites
Procedure: Scaling and root planing with solution — Mechanical instrumentation with sodium hypochlorite disinfective solution
  Arms: Scaling and root planing with solution

SUMMARY:
This study will determine whether the supplemental use of chemical pocket disinfection with scaling and root planing is more effective than scaling and root planing alone in clinically reducing periodontal probing depth (PD), reducing bleeding on probing (BOP), and gaining clinical attachment level (CAL). It also will assess whether chemical pocket disinfection with scaling and root planing will have an effect on biomarkers of inflammation.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the adjunctive use of chemical pocket disinfection with scaling and root planing is more effective than scaling and root planing alone in clinically reducing periodontal probing depth (PD), reducing bleeding on probing (BOP), and gaining clinical attachment level (CAL). It also will assess whether chemical pocket disinfection with scaling and root planing will have an effect on biomarkers of inflammation, as indicated by presence of pro- and anti-inflammatory cytokines, compared to scaling and root planing alone. The chemical pocket disinfection therapy consists of delivering a sodium hypochlorite solution followed by a neutralizing citric acid solution to the test site. Pro-inflammatory interleukin-1 beta and anti-inflammatory interleukin-1 receptor antagonist will be measured from the gingival crevicular fluid sampled from sites of interest.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal maintenance patients, have at least one pocket greater than or equal to 5 mm with bleeding on probing

Exclusion Criteria:

* Uncontrolled diabetics
* Regular users of nonsteroidal antiinflammatory drugs
* Individuals on anti-coagulants
* Individuals that have used antibiotics in the previous 3 months or require prophylactic antibiotic coverage
* Pregnant individuals

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
Probing depths | 3 months
  Periodontal probing depth (PD)

SECONDARY OUTCOMES:
Bleeding on probing | 3 months
  Incidence of bleeding during probing
Clinical attachment level | 3 months
  Clinical attachment level is calculated by adding gingival recession to probing depth; measures the connective tissue and epithelial attachment level relative to the cementoenamel junction
Inflammatory markers | 3 months
  Measure interleukin-1 beta and interleukin 1 receptor antagonist levels in gingival crevicular fluid from sites of interest

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Kaldahl, DDS, Study Director — UNMC College of Dentistry
Locations (1):
- UNMC College of Dentistry, Lincoln, Nebraska, United States